CLINICAL TRIAL: NCT03022253
Title: Liberal Versus Restrictive Platelet Transfusion for Treatment of Hemodynamically Significant Patent Ductus Arteriosus in Thrombocytopenic Preterm Neonates- A Randomized Open Label, Controlled Trial
Brief Title: Platelet Transfusion for Treatment of Patent Ductus Arteriosus in Thrombocytopenic Preterm Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sourabh Dutta, Dr, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2016/1090
Record Dates: First submitted 2016-06-25; First posted 2017-01-16 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Platelets
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; crocin; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal Platelet transfusion group (Experimental): Platelet transfusion to maintain a platelet count above 1,00,000 per microliter until one of the endpoints is met.
  As all subjects recruited in the trial will have hemodynamically significant (hs) PDA, they will all be medically treated as per standard of care. Treatment regimens will be as follows, depending on the discretion of the treating physician:
  Ibuprofen:
  Dosage-10 mg/kg stat followed by 5 mg/kg/dose x 2 doses at 24 hours intervals Route- oral
  Paracetamol:
  Dosage-15 mg/kg/dose every 6 hourly x 12 doses Route - IV
  Interventions: Biological: Liberal platelet transfusion; Drug: Paracetamol; Drug: Ibuprofen
- Restrictive platelet transfusion group (Active Comparator): Platelet transfusion for standard criteria.
  As all subjects recruited in the trial will have hemodynamically significant (hs) PDA, they will all be medically treated as per standard of care. Treatment regimens will be as follows, depending on the discretion of the treating physician:
  Ibuprofen:
  Dosage-10 mg/kg stat followed by 5 mg/kg/dose x 2 doses at 24 hours intervals Route- oral
  Paracetamol:
  Dosage-15 mg/kg/dose every 6 hourly x 12 doses Route - IV
  Interventions: Biological: Restrictive platelet transfusion; Drug: Paracetamol; Drug: Ibuprofen

INTERVENTIONS:
Biological: Liberal platelet transfusion — Liberal platelet transfusion: In Intervention group the investigators will transfuse platelet concentrates to maintain a platelet count above 1,00,000 per microliter until one of the following endpoints is met, whichever is applicable:
  1. PDA closes or
  2. A maximum of 120 hours after the point of randomisation
  Arms: Liberal Platelet transfusion group
Biological: Restrictive platelet transfusion — The investigators will transfuse platelets only if:
  (i) Platelet count is < 20,000 per microliter or (ii) Subject has a clinical bleed or (iii) Subject has platelet count < 50000 per microliter and requires a major non-neurosurgical interventional procedure as per the current standard of care, or (iv) Subject has a platelet count < 1, 00,000 per microliter and requires a neurosurgical procedure
  Arms: Restrictive platelet transfusion group
Drug: Paracetamol — As all subjects recruited in the trial will have hemodynamically significant (hs) PDA, they will all be medically treated as per standard of care. Treatment regimens will be as follows, depending on the discretion of the treating physician:
  Paracetamol:
  Dosage-15 mg/kg/dose every 6 hourly x 12 doses Route - IV
  Other Names: Crocin
Drug: Ibuprofen — As all subjects recruited in the trial will have hemodynamically significant (hs) PDA, they will all be medically treated as per standard of care. Treatment regimens will be as follows, depending on the discretion of the treating physician:
  Ibuprofen:
  Dosage-10 mg/kg stat followed by 5 mg/kg/dose x 2 doses at 24 hours intervals Route- oral
  Other Names: Brufen

SUMMARY:
Patent ductus arteriosus (PDA) is a common problem in preterm babies. Recently there have been various studies for and against an association between thrombocytopenia and PDA. A meta-analysis published in 2015 showed a marginally significant positive association between PDA and thrombocytopenia but these were all observational studies and there are no randomized controlled trials (RCT) on it. The investigators decided to conduct an RCT to determine whether liberal platelet transfusion criteria achieve earlier PDA closure rates than standard restrictive platelet transfusion criteria among thrombocytopenic preterm neonates (<35 weeks' gestation) with hemodynamically significant PDA presenting within the first 14 days of life. The investigators primary objective is to determine whether liberal platelet transfusion criteria achieve earlier PDA closure rates within 120 hours compared to standard restrictive platelet transfusion criteria among thrombocytopenic preterm neonates (<35 weeks' gestation) with hemodynamically significant PDA presenting within the first 14 days of life.

The investigators will stratify the study population based on platelet count, i.e < 50000 and 50000-100000 per microlitre, and will randomly allocate participants to control and intervention group. Babies in the intervention group will receive platelet transfusion to maintain the platelet count above 100,000 per microlitre. Babies in control group will receive platelets only when clinically indicated and as per current standard indications. The investigators will perform an echocardiogram at baseline to document a hemodynamically significant PDA (hsPDA) and then serially to look for the closure of PDA. Medical management of PDA will be as per unit policy. The investigators will follow the baby till PDA closes or 120 hours post randomization.

DETAILED DESCRIPTION:
Study Background:

Preterm babies are a unique group of patients in Newborn Intensive Care Unit. Patent ductus arteriosus (PDA) is a common complication related to the gestational age of preterm birth. In infants born at less than 32 weeks of gestation, the frequency of PDA has been reported from 50% to 80%. Physiologic ductus arteriosus closure occurs in the first 3 days after birth. The persistence of a PDA beyond the first postnatal days of life, however, is frequently associated with multiple severe complications, predominantly in the most immature infants It is currently believed that ductus arteriosus (DA) closure involves a two-step process. The first, 'provisional' closure is accomplished by smooth muscle cell contraction and ductus arteriosus (DA) constriction. Subsequently, the proliferation of cells within the former DA lumen leads to anatomical remodeling of the DA and permits permanent closure. Recently an association between the absolute platelet count and the closure of ductus arteriosus has been the focus of research. Various prospective and retrospective studies have been conducted for the same. In 2015 systematic review and meta-analysis by Sorina et al showed a significant positive association between PDA and thrombocytopenia. Hence the investigators planned randomized controlled trial to look for the effect of platelet transfusion on closure rates of ductus arteriosus.

Research question:

Do liberal platelet transfusion criteria achieve earlier PDA closure rates than standard restrictive platelet transfusion criteria among thrombocytopenic preterm neonates (<35 weeks gestation) with hemodynamically significant PDA presenting within the first 14 days of life?

Objectives:

Primary objective: To determine whether liberal platelet transfusion criteria achieve earlier PDA closure rates within 120 hours compared to standard restrictive platelet transfusion criteria among thrombocytopenic preterm neonates (<35 weeks gestation) with hemodynamically significant PDA presenting within the first 14 days of life.

Secondary objectives:

1. To determine the time period between platelet transfusion and closure of PDA.
2. To compare between the 2 groups:

   1. Proportion in whom PDA is open at 24 hours after the last dose of the course of medication
   2. Proportion in whom PDA is echocardiographically hemodynamically significant at 24 hours after the last dose of the course of medication
   3. Proportion in whom PDA is echocardiographically hemodynamically significant at 120 hours after randomization
   4. Cumulative volume of platelet concentrate received within 120 hours after randomization
   5. Any kind of clinical bleed within 120 hours after randomization
   6. New onset Intraventricular hemorrhage (IVH) of any grade within 120 hours after randomization
   7. New onset IVH of grade 3,4 within 120 hours after randomization
   8. Mortality within 120 hours after randomization
   9. Mortality anytime during hospital stay
   10. Duration of hospital stay
   11. Reopening rate of PDA that had initially closed within 120 hours of randomization

Study Design:

This will be a randomized, open-label, controlled trial.

Place of study Newborn unit of the Department of Pediatrics Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

Study period:

* Subject recruitment and data collection: January 2016 to December 2016 (12 months)
* Data analysis: January 2017 to March 2017 (3 months)
* Writing of dissertation: April 2017 to June 2017 (3 months)

Screening criteria (all must be fulfilled):

The investigators will screen all inborn and outborn neonates (admitted in Neonatal intensive care unit (NICU) or Neonatal nursery (NNN) for the following:

1. Gestational age up to 346/7 weeks
2. PDA detected for the first time at less than 14 days of postnatal age

Infants who meet the screening criteria will undergo an echocardiogram conducted by the 1st investigator and a platelet count and will be included if they fulfill all the following inclusion criteria mentioned below.

Procedure of platelet count:

The investigators will draw 0.5 ml of blood into an Ethylene diamine tetraacetic acid (EDTA) Container and immediately send it for analysis to the emergency lab Room No. 24 situated in Advanced Trauma Centre PGIMER Chandigarh. A technician will measure the platelet count by using an automated blood cell coulter (Sysmex KX-21 Coulter) situated in this lab. One of the co-investigators (N.V.) will ensure that the facility of platelet counts is available round-the-clock within a turnaround time of about 2 hours for subjects enrolled in the trial, and will also ensure quality control of the procedure.

Procedure of echocardiography:

The first investigator (JK) will perform the echocardiogram on a SonoSite MicroMaxx Portable Ultrasound Machine. Extremely low birth neonates (ELBW) neonates will be screened in first 48 hours as per unit policy, and the rest will undergo echocardiography only when there are clinical signs of PDA. Before performing the echocardiogram, the first investigator will use a website-generated unique, random code number as the patient identifier. The first investigator will take a backup of each echocardiogram immediately on an external hard drive and the video files will be named with the same website-generated random code number. One of the co-investigators (VS or SS) will review the code numbered echocardiograms. VS and SS will be masked to the identity and clinical details of the patients. The key to the code numbers will be maintained by JK and Sourabh Dutta (SD). The echocardiographic diagnosis of PDA by VS or SS will be considered to be the gold standard.

The following information will be recorded for each echocardiogram:

1. Whether the ductus arteriosus is patent or closed.
2. If it is patent, Transductal diameter, Ductal velocity, Antegrade left PA diastolic flow, Left Atrium/Aorta (LA/Ao) ratio, E/A, Isovolumic relaxation time (IVRT) , Absent or reversed diastolic blood flow pattern in descending thoracic aorta.

Patient information and informed consent:

The 1st investigator (J.K.) will approach parents of subjects that meet the above eligibility criteria for possible enrollment in the study. The first investigator will provide them a detailed information sheet and also give a verbal explanation about the study. The first investigator will enroll neonates only after obtaining written informed consent from one of the parents.

Baseline data:

The investigators will record baseline maternal and neonatal data.

Medical treatment of PDA:

As all subjects recruited in the trial will have hemodynamically significant PDA, they will all be medically treated. Details are given under intervention heading.

Some subjects may be recruited in another ongoing RCT during the initial months of this trial. The other RCT compares paracetamol and ibuprofen in a blinded fashion amongst subjects with hemodynamically significant PDA for the closure of PDA. For such subjects, the trial drug regime will be followed. The index trial will not be affected by being co-recruited in the other ongoing RCT. If a particular dose of medication cannot be given because of a contraindication (an adverse effect or adverse clinical condition) that arises during the course of treatment, that dose will be deferred until it is safe to administer the dose. The duration of medical treatment will be taken as the total duration inclusive of the deferred dose/s.

Randomization:

The investigators will allocate patients according to a stratified, block randomised design. The investigators will stratify patients into the following strata: a) platelet count < 50,000 per microliter b) platelet count 50,000-100,000 per microliter. The Chief guide Sourabh Dutta (S.D.) will generate the randomisation sequence and construct randomly varying, permuted, even-numbered blocks for each stratum. The chief guide will conceal the block sizes until the end of the study. Each stratum will have its independent randomisation sequence. After the 1st investigator identifies the stratum, S.D. will randomly allocate subjects to an intervention or control group. The investigators will ensure concealment of allocation by using serially numbered opaque sealed envelopes which will bear a slip of paper with the allocation group.

Allocation groups:

Intervention group: The investigators will transfuse platelet concentrates to maintain platelet count above 1, 00,000 per microliter (details are given under Arms and Intervention) The investigators will aggressively monitor platelet counts in the intervention group, depending upon the stratum in which the subject is enrolled.

In the stratum that has a baseline platelet count less than 50,000 per microliter, there is very little chance that the platelet count will rise to more than 100,000 per microliter with a single platelet concentrate transfusion. In this stratum, two back to back platelet concentrates (20 ml/kg each) will be transfused without performing a platelet count in between the 2 tests transfusions.

In the stratum that has a baseline platelet count from 50,000 to 100,000 per microliter, a platelet count will be performed after a single transfusion.

In both strata, platelet count will be repeated in a window period of 2 hours after the end of the platelet transfusion. The investigators will attempt to club this platelet count with another blood sampling for clinical indications if possible. The investigators will attempt to get the post-transfusion platelet count within a turnaround time of 2 hours. If the subject has a platelet count less than 100,000 per microliter, the investigators will repeat a platelet transfusion, and so on, subject to a maximum volume of 40 ml/kg/day of platelet concentrates in a 24-hour period (defined as 8 AM to 8 AM next day). The investigators will temporarily stop transfusing platelet concentrates once the investigators get a value of above 100,000 per microliter. In addition to the platelet counts performed post-transfusion, the investigators will also perform platelet counts for the following indications:

(i) Clinical bleeds (ii) A routine platelet count once in every 24 hours until PDA closes or the criterion of 120 hours post randomization is met.

The platelet count for clinical bleeds and routine platelet counts will not be repeated in case a platelet count post-transfusion is already available within a window period of 4 hours prior.

Control group: (details are given under Arms and Intervention) In the control group, the investigators will perform platelet counts as per the standard unit practices. A platelet count will be repeated whenever the subject is next sampled for a clinical indication or a longer with routine samples in the evening or morning. A platelet transfusion will be repeated if the platelet count falls to less than 20,000 per microliter or if any of the above criteria are met.

In both groups, platelet concentrates will be transfused according to platelet count prior to transfusion. In babies with platelet count < 50000, 50-75000 and 75-1, 00, 00 per microliter the investigators will transfuse @ 20, 15 and 10 ml/kg/transfusion respectively up to a maximum of 40 ml/kg/day. The investigators will administer injection furosemide 0.5 mg/kg as slow IV injection midway through the transfusion if the treating team clinically feels that the patient is likely to develop congestive cardiac failure or pulmonary edema.

Study endpoints:

Subjects will be followed up in the study until the earliest among

1. Withdrawal of consent
2. Discharge from hospital
3. Death

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age up to 34 6/7 weeks
2. PDA detected for the first time at less than 14 days of postnatal age
3. Clinically and/or echocardiographically hemodynamically significant PDA Note: ELBW neonates will be screened in first 48 hours as per unit policy; the rest will undergo echocardiography only when there are clinical signs of PDA.
4. Platelet count within 24 hours prior to inclusion is less than 100,000 per microliter.

Note: If a platelet count is already available within 24 hours prior to inclusion it will be accepted as a valid platelet count. If not, an urgent absolute platelet count will be performed.

Exclusion Criteria:

1. Echocardiographically proven structural congenital heart disease.
2. Major life-threatening malformation
3. Received platelet concentrate between the last available platelet count and the point of randomisation

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Time to closure of PDA post randomization | within 120 hours post randomisation
  Time point at which closure (Absence of flow in PDA on colour doppler) is documented first time will be considered as time to closure of PDA

SECONDARY OUTCOMES:
Proportion of participants in whom PDA is open | at 120 hours after randomization
  PDA will be considered open if there is presence of flow on colour doppler
Proportion of participants in whom PDA is echocardiographically hemodynamically significant | at 120 hours after randomization
  hemodynamic significance is defined somewhere else in text
Cumulative volume of platelet concentrate received | within 120 hours after randomization
  Total volume in ml/kg will be recorded
Number of participants with Clinical bleed of any kind ( defined below) | within 120 hours after randomization
  Any visible fresh oral, nasal, endotracheal, gastrointestinal or skin bleed will be considered as clinical bleed.
New onset IVH of any grade | within 120 hours after randomization
  Cranial ultrasound will be done as per protocol to look for IVH
New onset IVH of grade 3or 4 | within 120 hours after randomization
  Cranial ultrasound will be done as per protocol to look for IVH
Mortality | within 120 hours after randomization
  It stands for all cause mortality
Mortality | All subjects will be part of the study until death or discharge from the hospital. Timeframe for measuring mortality as an outcome is from the point of randomisation through the study period which will be approximately upto 30 days post randomisation
  It stands for all cause mortality
Duration of hospital stay | All subjects will be part of the study until death or discharge from the hospital.Timeframe for measuring duration of hospital stay is from the point of randomisation through the study period which will be approximately upto 30 days post randomisation
  Duration of stay will be from date of birth to date of discharge/referral or death
Reopening rate of PDA that had initially closed | within 120 hours of randomization
  It will include situation where PDA closure was documented on two consecutive occasions 24 hours apart and then at later stage it opens.

CONTACTS AND LOCATIONS:
Overall Officials: Sourabh Dutta, MD, Study Director — Post Graduate Institute of Medical Education and Research; Chandigarh, India
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bancalari E, Claure N, Gonzalez A. Patent ductus arteriosus and respiratory outcome in premature infants. Biol Neonate. 2005;88(3):192-201. doi: 10.1159/000087582. PMID 16210841
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Adrouche-Amrani L, Green RS, Gluck KM, Lin J. Failure of a repeat course of cyclooxygenase inhibitor to close a PDA is a risk factor for developing chronic lung disease in ELBW infants. BMC Pediatr. 2012 Jan 27;12:10. doi: 10.1186/1471-2431-12-10. PMID 22284694
- [Background] Echtler K, Stark K, Lorenz M, Kerstan S, Walch A, Jennen L, Rudelius M, Seidl S, Kremmer E, Emambokus NR, von Bruehl ML, Frampton J, Isermann B, Genzel-Boroviczeny O, Schreiber C, Mehilli J, Kastrati A, Schwaiger M, Shivdasani RA, Massberg S. Platelets contribute to postnatal occlusion of the ductus arteriosus. Nat Med. 2010 Jan;16(1):75-82. doi: 10.1038/nm.2060. Epub 2009 Dec 6. PMID 19966813
- [Background] Simon SR, van Zogchel L, Bas-Suarez MP, Cavallaro G, Clyman RI, Villamor E. Platelet Counts and Patent Ductus Arteriosus in Preterm Infants: A Systematic Review and Meta-Analysis. Neonatology. 2015;108(2):143-51. doi: 10.1159/000431281. Epub 2015 Jul 7. PMID 26159239
- [Background] Stoller JZ, Demauro SB, Dagle JM, Reese J. Current Perspectives on Pathobiology of the Ductus Arteriosus. J Clin Exp Cardiolog. 2012 Jun 15;8(1):S8-001. doi: 10.4172/2155-9880.S8-001. PMID 23519783
- [Background] Loftin CD, Trivedi DB, Tiano HF, Clark JA, Lee CA, Epstein JA, Morham SG, Breyer MD, Nguyen M, Hawkins BM, Goulet JL, Smithies O, Koller BH, Langenbach R. Failure of ductus arteriosus closure and remodeling in neonatal mice deficient in cyclooxygenase-1 and cyclooxygenase-2. Proc Natl Acad Sci U S A. 2001 Jan 30;98(3):1059-64. doi: 10.1073/pnas.98.3.1059. Epub 2001 Jan 23. PMID 11158594
- [Background] Yu Y, Funk CD. A novel genetic model of selective COX-2 inhibition: comparison with COX-2 null mice. Prostaglandins Other Lipid Mediat. 2007 Jan;82(1-4):77-84. doi: 10.1016/j.prostaglandins.2006.05.021. Epub 2006 Jul 7. PMID 17164135
- [Background] Reese J, Paria BC, Brown N, Zhao X, Morrow JD, Dey SK. Coordinated regulation of fetal and maternal prostaglandins directs successful birth and postnatal adaptation in the mouse. Proc Natl Acad Sci U S A. 2000 Aug 15;97(17):9759-64. doi: 10.1073/pnas.97.17.9759. PMID 10944235
- [Background] Reese J, Waleh N, Poole SD, Brown N, Roman C, Clyman RI. Chronic in utero cyclooxygenase inhibition alters PGE2-regulated ductus arteriosus contractile pathways and prevents postnatal closure. Pediatr Res. 2009 Aug;66(2):155-61. doi: 10.1203/PDR.0b013e3181aa07eb. PMID 19390487
- [Background] Derzbach L, Treszl A, Balogh A, Vasarhelyi B, Tulassay T, Rigo J J. Gender dependent association between perinatal morbidity and estrogen receptor-alpha Pvull polymorphism. J Perinat Med. 2005;33(5):461-2. doi: 10.1515/JPM.2005.082. PMID 16238543
- [Background] Bokodi G, Derzbach L, Banyasz I, Tulassay T, Vasarhelyi B. Association of interferon gamma T+874A and interleukin 12 p40 promoter CTCTAA/GC polymorphism with the need for respiratory support and perinatal complications in low birthweight neonates. Arch Dis Child Fetal Neonatal Ed. 2007 Jan;92(1):F25-9. doi: 10.1136/adc.2005.086421. Epub 2006 Jun 5. PMID 16754651
- [Background] Gonzalez A, Sosenko IR, Chandar J, Hummler H, Claure N, Bancalari E. Influence of infection on patent ductus arteriosus and chronic lung disease in premature infants weighing 1000 grams or less. J Pediatr. 1996 Apr;128(4):470-8. doi: 10.1016/s0022-3476(96)70356-6. PMID 8618179
- [Background] Rojas MA, Gonzalez A, Bancalari E, Claure N, Poole C, Silva-Neto G. Changing trends in the epidemiology and pathogenesis of neonatal chronic lung disease. J Pediatr. 1995 Apr;126(4):605-10. doi: 10.1016/s0022-3476(95)70362-4. PMID 7699543
- [Background] Waleh N, Hodnick R, Jhaveri N, McConaghy S, Dagle J, Seidner S, McCurnin D, Murray JC, Ohls R, Clyman RI. Patterns of gene expression in the ductus arteriosus are related to environmental and genetic risk factors for persistent ductus patency. Pediatr Res. 2010 Oct;68(4):292-7. doi: 10.1203/PDR.0b013e3181ed8609. PMID 20581741
- [Background] BORN GV, DAWES GS, MOTT JC, RENNICK BR. The constriction of the ductus arteriosus caused by oxygen and by asphyxia in newborn lambs. J Physiol. 1956 May 28;132(2):304-42. doi: 10.1113/jphysiol.1956.sp005526. No abstract available. PMID 13320399
- [Background] KOVALCIK V. THE RESPONSE OF THE ISOLATED DUCTUS ARTERIOSUS TO OXYGEN AND ANOXIA. J Physiol. 1963 Nov;169(1):185-97. doi: 10.1113/jphysiol.1963.sp007249. No abstract available. PMID 14078057
- [Background] MOSS AJ, EMMANOUILIDES GC, ADAMS FH, CHUANG K. RESPONSE OF DUCTUS ARTERIOSUS AND PULMONARY AND SYSTEMIC ARTERIAL PRESSURE TO CHANGES IN OXYGEN ENVIRONMENT IN NEWBORN INFANTS. Pediatrics. 1964 Jun;33:937-44. No abstract available. PMID 14169640
- [Background] Fay FS. Guinea pig ductus arteriosus. I. Cellular and metabolic basis for oxygen sensitivity. Am J Physiol. 1971 Aug;221(2):470-9. doi: 10.1152/ajplegacy.1971.221.2.470. No abstract available. PMID 5560296
- [Background] Smith GC. The pharmacology of the ductus arteriosus. Pharmacol Rev. 1998 Mar;50(1):35-58. No abstract available. PMID 9549757
- [Background] Ward JP. Oxygen sensors in context. Biochim Biophys Acta. 2008 Jan;1777(1):1-14. doi: 10.1016/j.bbabio.2007.10.010. Epub 2007 Nov 1. PMID 18036551
- [Background] Fleming I. Vascular cytochrome p450 enzymes: physiology and pathophysiology. Trends Cardiovasc Med. 2008 Jan;18(1):20-5. doi: 10.1016/j.tcm.2007.11.002. PMID 18206805
- [Background] Baragatti B, Schwartzman ML, Angeloni D, Scebba F, Ciofini E, Sodini D, Ottaviano V, Nencioni S, Paolicchi A, Graves JP, Zeldin DC, Gotlinger K, Luin S, Coceani F. EDHF function in the ductus arteriosus: evidence against involvement of epoxyeicosatrienoic acids and 12S-hydroxyeicosatetraenoic acid. Am J Physiol Heart Circ Physiol. 2009 Dec;297(6):H2161-8. doi: 10.1152/ajpheart.00576.2009. Epub 2009 Oct 2. PMID 19801493
- [Background] Roulet MJ, Coburn RF. Oxygen-induced contraction in the guinea pig neonatal ductus arteriosus. Circ Res. 1981 Oct;49(4):997-1002. doi: 10.1161/01.res.49.4.997. PMID 7273368
- [Background] Nakanishi T, Gu H, Hagiwara N, Momma K. Mechanisms of oxygen-induced contraction of ductus arteriosus isolated from the fetal rabbit. Circ Res. 1993 Jun;72(6):1218-28. doi: 10.1161/01.res.72.6.1218. PMID 8495551
- [Background] Tristani-Firouzi M, Reeve HL, Tolarova S, Weir EK, Archer SL. Oxygen-induced constriction of rabbit ductus arteriosus occurs via inhibition of a 4-aminopyridine-, voltage-sensitive potassium channel. J Clin Invest. 1996 Nov 1;98(9):1959-65. doi: 10.1172/JCI118999. PMID 8903313
- [Background] Weir EK, Lopez-Barneo J, Buckler KJ, Archer SL. Acute oxygen-sensing mechanisms. N Engl J Med. 2005 Nov 10;353(19):2042-55. doi: 10.1056/NEJMra050002. No abstract available. PMID 16282179
- [Background] Michelakis E, Rebeyka I, Bateson J, Olley P, Puttagunta L, Archer S. Voltage-gated potassium channels in human ductus arteriosus. Lancet. 2000 Jul 8;356(9224):134-7. doi: 10.1016/S0140-6736(00)02452-1. PMID 10963252
- [Background] Archer SL, Wu XC, Thebaud B, Moudgil R, Hashimoto K, Michelakis ED. O2 sensing in the human ductus arteriosus: redox-sensitive K+ channels are regulated by mitochondria-derived hydrogen peroxide. Biol Chem. 2004 Mar-Apr;385(3-4):205-16. doi: 10.1515/BC.2004.014. PMID 15134333
- [Background] Arcilla RA, Thilenius OG, Ranniger K. Congestive heart failure from suspected ductal closure in utero. J Pediatr. 1969 Jul;75(1):74-8. doi: 10.1016/s0022-3476(69)80103-4. PMID 4239830
- [Background] Zuckerman H, Reiss U, Rubinstein I. Inhibition of human premature labor by indomethacin. Obstet Gynecol. 1974 Dec;44(6):787-92. No abstract available. PMID 4437814
- [Background] Coceani F, Olley PM. The response of the ductus arteriosus to prostaglandins. Can J Physiol Pharmacol. 1973 Mar;51(3):220-5. doi: 10.1139/y73-031. No abstract available. PMID 4705142
- [Background] Coceani F, Olley PM, Bodach E. Lamb ductus arteriosus: effect of prostaglandin synthesis inhibitors on the muscle tone and the response to prostaglandin E2. Prostaglandins. 1975 Feb;9(2):299-308. doi: 10.1016/0090-6980(75)90034-9. PMID 1135442
- [Background] Sharpe GL, Thalme B, Larsson KS. Studies on closure of the ductus arteriosus. XI. Ductal closure in utero by a prostaglandin synthetase inhibitor. Prostaglandins. 1974 Dec 10;8(5):363-8. doi: 10.1016/0090-6980(74)90110-5. No abstract available. PMID 4453621
- [Background] Starling MB, Elliott RB. The effects of prostaglandins, prostaglandin inhibitors, and oxygen on the closure of the ductus arteriosus, pulmonary arteries and umbilical vessels in vitro. Prostaglandins. 1974 Nov 10;8(3):187-203. doi: 10.1016/0090-6980(74)90042-2. No abstract available. PMID 4215100
- [Background] Friedman WF, Hirschklau MJ, Printz MP, Pitlick PT, Kirkpatrick SE. Pharmacologic closure of patent ductus arteriosus in the premature infant. N Engl J Med. 1976 Sep 2;295(10):526-9. doi: 10.1056/NEJM197609022951003. PMID 820994
- [Background] Heymann MA, Rudolph AM, Silverman NH. Closure of the ductus arteriosus in premature infants by inhibition of prostaglandin synthesis. N Engl J Med. 1976 Sep 2;295(10):530-3. doi: 10.1056/NEJM197609022951004. PMID 950959
- [Background] Coceani F, Olley PM, Bishai I, Bodach E, Heaton J, Nashat M, White E. Prostaglandins and the control of muscle tone in the ductus arteriosus. Adv Exp Med Biol. 1977;78:135-42. doi: 10.1007/978-1-4615-9035-4_10. PMID 899912
- [Background] Coceani F, White E, Bodach E, Olley PM. Age-dependent changes in the response of the lamb ductus arteriosus to oxygen and ibuprofen. Can J Physiol Pharmacol. 1979 Aug;57(8):825-31. doi: 10.1139/y79-126. PMID 497895
- [Background] Schneider DJ, Moore JW. Patent ductus arteriosus. Circulation. 2006 Oct 24;114(17):1873-82. doi: 10.1161/CIRCULATIONAHA.105.592063. No abstract available. PMID 17060397
- [Background] Clyman RI, Chan CY, Mauray F, Chen YQ, Cox W, Seidner SR, Lord EM, Weiss H, Waleh N, Evans SM, Koch CJ. Permanent anatomic closure of the ductus arteriosus in newborn baboons: the roles of postnatal constriction, hypoxia, and gestation. Pediatr Res. 1999 Jan;45(1):19-29. doi: 10.1203/00006450-199901000-00005. PMID 9890604
- [Background] Keck M, Resnik E, Linden B, Anderson F, Sukovich DJ, Herron J, Cornfield DN. Oxygen increases ductus arteriosus smooth muscle cytosolic calcium via release of calcium from inositol triphosphate-sensitive stores. Am J Physiol Lung Cell Mol Physiol. 2005 May;288(5):L917-23. doi: 10.1152/ajplung.00403.2004. Epub 2005 Feb 4. PMID 15695541
- [Background] Weir EK, Obreztchikova M, Vargese A, Cabrera JA, Peterson DA, Hong Z. Mechanisms of oxygen sensing: a key to therapy of pulmonary hypertension and patent ductus arteriosus. Br J Pharmacol. 2008 Oct;155(3):300-7. doi: 10.1038/bjp.2008.291. Epub 2008 Jul 21. PMID 18641675
- [Background] Thebaud B, Michelakis ED, Wu XC, Moudgil R, Kuzyk M, Dyck JR, Harry G, Hashimoto K, Haromy A, Rebeyka I, Archer SL. Oxygen-sensitive Kv channel gene transfer confers oxygen responsiveness to preterm rabbit and remodeled human ductus arteriosus: implications for infants with patent ductus arteriosus. Circulation. 2004 Sep 14;110(11):1372-9. doi: 10.1161/01.CIR.0000141292.28616.65. Epub 2004 Sep 7. PMID 15353504
- [Background] Thebaud B, Wu XC, Kajimoto H, Bonnet S, Hashimoto K, Michelakis ED, Archer SL. Developmental absence of the O2 sensitivity of L-type calcium channels in preterm ductus arteriosus smooth muscle cells impairs O2 constriction contributing to patent ductus arteriosus. Pediatr Res. 2008 Feb;63(2):176-81. doi: 10.1203/PDR.0b013e31815ed059. PMID 18091358
- [Background] Kajimoto H, Hashimoto K, Bonnet SN, Haromy A, Harry G, Moudgil R, Nakanishi T, Rebeyka I, Thebaud B, Michelakis ED, Archer SL. Oxygen activates the Rho/Rho-kinase pathway and induces RhoB and ROCK-1 expression in human and rabbit ductus arteriosus by increasing mitochondria-derived reactive oxygen species: a newly recognized mechanism for sustaining ductal constriction. Circulation. 2007 Apr 3;115(13):1777-88. doi: 10.1161/CIRCULATIONAHA.106.649566. Epub 2007 Mar 12. PMID 17353442
- [Background] Hong Z, Hong F, Olschewski A, Cabrera JA, Varghese A, Nelson DP, Weir EK. Role of store-operated calcium channels and calcium sensitization in normoxic contraction of the ductus arteriosus. Circulation. 2006 Sep 26;114(13):1372-9. doi: 10.1161/CIRCULATIONAHA.106.641126. Epub 2006 Sep 18. PMID 16982938
- [Background] Coceani F, Kelsey L. Endothelin-1 release from lamb ductus arteriosus: relevance to postnatal closure of the vessel. Can J Physiol Pharmacol. 1991 Feb;69(2):218-21. doi: 10.1139/y91-033. PMID 2054736
- [Background] Fineman JR, Takahashi Y, Roman C, Clyman RI. Endothelin-receptor blockade does not alter closure of the ductus arteriosus. Am J Physiol. 1998 Nov;275(5):H1620-6. doi: 10.1152/ajpheart.1998.275.5.H1620. PMID 9815069
- [Background] Weiss H, Cooper B, Brook M, Schlueter M, Clyman R. Factors determining reopening of the ductus arteriosus after successful clinical closure with indomethacin. J Pediatr. 1995 Sep;127(3):466-71. doi: 10.1016/s0022-3476(95)70084-6. PMID 7658282
- [Background] Fujioka K, Morioka I, Miwa A, Morikawa S, Shibata A, Yokoyama N, Matsuo M. Does thrombocytopenia contribute to patent ductus arteriosus? Nat Med. 2011 Jan;17(1):29-30; author reply 30-1. doi: 10.1038/nm0111-29. No abstract available. PMID 21217670
- [Background] Shah NA, Hills NK, Waleh N, McCurnin D, Seidner S, Chemtob S, Clyman R. Relationship between circulating platelet counts and ductus arteriosus patency after indomethacin treatment. J Pediatr. 2011 Jun;158(6):919-923.e1-2. doi: 10.1016/j.jpeds.2010.11.018. Epub 2010 Dec 30. PMID 21195414
- [Background] Alyamac Dizdar E, Ozdemir R, Sari FN, Yurttutan S, Gokmen T, Erdeve O, Emre Canpolat F, Uras N, Suna Oguz S, Dilmen U. Low platelet count is associated with ductus arteriosus patency in preterm newborns. Early Hum Dev. 2012 Oct;88(10):813-6. doi: 10.1016/j.earlhumdev.2012.05.007. Epub 2012 Jun 18. PMID 22717423
- [Background] Sallmon H, Weber SC, Huning B, Stein A, Horn PA, Metze BC, Dame C, Buhrer C, Felderhoff-Muser U, Hansmann G, Koehne P. Thrombocytopenia in the first 24 hours after birth and incidence of patent ductus arteriosus. Pediatrics. 2012 Sep;130(3):e623-30. doi: 10.1542/peds.2012-0499. Epub 2012 Aug 6. PMID 22869835
- [Background] Bas-Suarez MP, Gonzalez-Luis GE, Saavedra P, Villamor E. Platelet counts in the first seven days of life and patent ductus arteriosus in preterm very low-birth-weight infants. Neonatology. 2014;106(3):188-94. doi: 10.1159/000362432. Epub 2014 Jul 5. PMID 25012267
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Ohlsson A, Walia R, Shah SS. Ibuprofen for the treatment of patent ductus arteriosus in preterm and/or low birth weight infants. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD003481. doi: 10.1002/14651858.CD003481.pub5. PMID 23633310
- [Background] O'Riordan JM, Fitzgerald J, Smith OP, Bonnar J, Gorman WA; National Blood Users Group. Transfusion of blood components to infants under four months: review and guidelines. Ir Med J. 2007 Jun;100(6):suppl 1-24 following 496. No abstract available. PMID 17668683
- [Derived] Kumar J, Dutta S, Sundaram V, Saini SS, Sharma RR, Varma N. Platelet Transfusion for PDA Closure in Preterm Infants: A Randomized Controlled Trial. Pediatrics. 2019 May;143(5):e20182565. doi: 10.1542/peds.2018-2565. Epub 2019 Apr 2. PMID 30940676